CLINICAL TRIAL: NCT06784401
Title: Oncologic and Functional Outcome and Quality of Life in Patients Treated for Laryngeal Cancer. (Original Title in Italian Language: "Il Trattamento Del Carcinoma Laringeo: Outcome Oncologico, Funzionale e Quality of Life")
Brief Title: Oncologic and Functional Outcome and Quality of Life in Patients Treated for Laryngeal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: LARYNX2023
Record Dates: First submitted 2024-11-28; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-01

CONDITIONS: Laryngeal Cancer
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about oncologic and functional outcome and investigate quality of life in patients treated for laryngeal cancer.

DETAILED DESCRIPTION:
Adult (>=18 years of age) patients treated by surgery and/or radiation therapy are enrolled retrospectively.

The main question it aims to answer is:

Is voice after total laryngectomy with voice prosthesis better than voice after open partial horizzontal laryngectomy? Subjective and objective scales and parameters are used.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for laryngeal cancer diagnosed by histopathologic examination

Exclusion Criteria:

* Patients lost at follow up
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (>= 18 years) of both sexes treated and followed for laryngeal cancer at the Department of Otollaryngology and Audiology of the University Hospital of Bologna.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-02 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Oncologic and functional outcome in patients treated for laryngeal cancer. | through study completion, an average of 1 year
  Compare the functional phonatory outcome assessed through objective parameters and subjective scales (GRBAS scale and INFVo Visual Analogue rating Scales) in patients undergoing total laryngectomy with placement of phonatory prosthesis with patients undergoing partial laryngectomy.
  Compare the functional phonatory outcome assessed by objective parameters and subjective scales (GRBAS scale and INFVo Visual Analogue rating Scales) in patients undergoing microlaryngoscopy cordectomy with patients undergoing exclusive radiotherapy for glottic cancer.
  Identify and describe phonation patterns in patients undergoing laryngectomy partial laryngectomy, evaluating possible associations between phonation patterns and phonatory outcomes.

SECONDARY OUTCOMES:
Quality of life in patients treated for laryngeal cancer. | through study completion, an average of 1 year
  To compare the quality of life and voice rate of satisfaction by subjective questionnaires (Voice Handicap Index - 10 and I-SECEL) in patients undergoing the different surgical techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Botti, MD, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy